CLINICAL TRIAL: NCT00790166
Title: Effects of nCPAP With and Without Humidification on: Inspiratory Temperature, Humidity, Saccharine Transit Time, Nasal Lavage and in Vitro Mucus Properties in Patients With Obstructive Sleep Apnea
Brief Title: Effects of Humidity (During CPAP Treatment) on Mucociliary Clearance in Patients With Obstructive Sleep Apnea
Acronym: CIA-6
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OSA CPAP,ThemoSmartMCC, Brasil
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2009-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- CPAP + ThermoSmart™ humidity (Active Comparator)
  Interventions: Device: CPAP + ThermoSmart™ humidity
- CPAP + Conventional humidity (Active Comparator)
  Interventions: Device: CPAP + Conventional humidity
- CPAP + No added humidity (Active Comparator)
  Interventions: Device: CPAP + No added humidity

INTERVENTIONS:
Device: CPAP + ThermoSmart™ humidity — an absolute humidity (AH) of 28 mg/l +/- 2mg/l
  Arms: CPAP + ThermoSmart™ humidity
Device: CPAP + Conventional humidity — an absolute humidity (AH) of 18 mg/l +/- 2 mg/l
  Arms: CPAP + Conventional humidity
Device: CPAP + No added humidity — ambient humidity
  Arms: CPAP + No added humidity

SUMMARY:
That the level of humidification delivered to patients during CPAP treatment will alter the subjects mucociliary clearance rate and related mucus properties.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe obstructive sleep apnea - Apnea Hypopnea Index (AHI) > 15
* 75% of events during the diagnostic study must be obstructive

Exclusion Criteria:

* Currently using CPAP treatment OR have used it in the past 4 weeks
* Intolerance of CPAP and/or CPAP mask in the past or during the titration night
* Mouth breather (unable to breath through mouth for the study period)
* < 18years old
* Nasal CPAP intolerance determined in the PSG-CPAP titration study
* Serious nasal issues
* Acute upper airway disease
* Smoker
* COPD
* Congestive heart failure
* Neuromuscular disease
* Stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06-24 (Actual); Study Completion 2009-06-24 (Actual)

PRIMARY OUTCOMES:
mucociliary clearance. | pre and post cpap treatment with varying levels of humidity

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi, MD, Principal Investigator — Faculty of Medicine: Pulmonology: University of Sao Paulo Hospital
Locations (1):
- Faculty of Medicine: Pulmonology: University of Sao Paulo Hospital, São Paulo, Brazil